CLINICAL TRIAL: NCT07129304
Title: Design And Analysis of The Effectiveness of Collaborative Virtual Reality Environment Versus Non-Immersive Virtual Reality in the Rehabilitation of Patients With Parkinson's Disease
Brief Title: Design And Analysis of The Effectiveness of CVRE VS Non-Immersive VR in the Rehabilitation of Parkinson
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Superior University (Other)
Responsible Party: Principal Investigator, Muhammad Naveed Babur, Principal Investigator, Superior University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Health Services Research
Other Study IDs: PhDRSW/Batch-Fall23/2227
Record Dates: First submitted 2025-08-12; First posted 2025-08-19 (Actual); Last update posted 2025-08-19 (Actual); Status verified 2025-08

CONDITIONS: Parkinson Disease
MeSH Terms: conditions — Parkinson Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Collaborative Virtual Reality with Routine Physical Therapy (Experimental)
  Interventions: Combination Product: Collaborative Virtual Reality with Routine Physical Therapy
- Non-Immersive Virtual Reality with Routine Physical Therapy (Experimental)
  Interventions: Combination Product: Non-Immersive Virtual Reality with Routine Physical Therapy

INTERVENTIONS:
Combination Product: Collaborative Virtual Reality with Routine Physical Therapy — patients will receive routine Physiotherapy treatment and additional treatment in a Collaborative Virtual Reality Environment for 30 minutes per session 3 times /week for minimum of 8 weeks. There will be a real time interaction in this group between patients and Physiotherapist in the virtual environment. The tasks in the CVE will focus on motor control, balance, coordination, and social engagement while routine Physical Therapy session will consist of performing exercises based on similar goals of improving motor skills, enhanced coordination, functional mobility, muscle strength and stretching exercises.
  Arms: Collaborative Virtual Reality with Routine Physical Therapy
Combination Product: Non-Immersive Virtual Reality with Routine Physical Therapy — Patients will receive routine physiotherapy treatment along with the engagement with computer-based virtual rehabilitation content displayed on a standard computer monitor/ LED screen. There will be no real time interaction in this group between patients and Physiotherapist in the virtual environment. Patients will be viewing pre-recorded videos of therapeutic exercises, demonstration, and / or on-screen instructions and cues for performing exercises. This group's patients will be treated with non- immersive virtual reality along with routine physical therapy for 30 minutes session 3 times /week for 8 weeks. Routine Physical Therapy session will consist of performing exercise based on the goal of improving motor skills, enhanced coordination, posture correction, gait efficiency, functional mobility, muscle strength and endurance training, stretching exercises where required.
  Arms: Non-Immersive Virtual Reality with Routine Physical Therapy

SUMMARY:
This study is being conducted to investigate the effect of Collaborative Virtual Reality Environments versus non-immersive Virtual reality-based rehabilitation in addition to the conventional Physical Therapy for patients with Parkinson's Disease to improve the motor, cognitive function, and overall quality of life.

DETAILED DESCRIPTION:
Parkinson's Disease is a progressive, neurodegenerative disorder with sign and symptoms of resting tremor, rigidity, retropulsion, stooping posture, sluggishness of spontaneous actions, with masked face. Parkinson's disease is increasing worldwide every year. Besides medical or surgical treatment, task-oriented Physical Therapy exercises have shown improvement in balance, reducing falls, and enhancing motor functions. Virtual reality (VR) has also appeared to be a promising means for rehabilitation in this disease. Collaborative Virtual Environments are shared digital spaces that enable real-time collaboration and interaction, often represented through avatars. Rehabilitation treatment with such advanced virtual reality technology i.e., comparing Collaborative Virtual Environments (CVEs) and Non-Immersive Virtual Reality to enhance motor functions along with cognitive tasks in Parkinson's disease may transform Physiotherapy rehabilitation by advocating engaging, effective, and scalable interventions, ultimately improving the outcomes and quality of life in Parkinson's disease.

ELIGIBILITY:
Inclusion Criteria:

* Gender: Both Male and Female genders patients
* Age Range: 40 years -80 Years
* Diagnosis: Clinically diagnosed patients of idiopathic Parkinson Disease classified as mild to moderate severity according to the modified Hoehn & Yahr stages I-III.
* Cognitive Function: Adequate cognitive function as assessed by Mini Mental State Examination (score ≥ 24)
* Functional Ability: can walk independently, must have sufficient physical and cognitive ability to engage in virtual rehabilitation sessions.

Exclusion Criteria:

* History of any neurological conditions other than Parkinson's disease.
* History of visual auditory, or motor impairments unrelated to Parkinson's Disease.
* History of orthopedic injury leading to complications like any deformity.
* Diagnosed phobia of virtual environment.
* Comorbidities that hinder participation in the treatment (e.g., advanced dementia).
* Patient taking another medication affecting neurological condition.

Ages: 40 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 60 (Actual)
Dates: Start 2025-04-17 (Actual); Primary Completion 2026-04-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Unified Parkinson's disease Rating Scale Part III | 24 Months
  The UPDRS Part III is a tool frequently employed in clinical settings to assess the motor functions of individuals with Parkinson's Disease. It encompasses a series of 31 items, which specifically evaluate motor symptoms such as tremor, rigidity, bradykinesia (slowness of movement), postural instability, and other related motor impairments.
  • Scoring: Total score range: 0 to 199. Higher scores indicate more severe motor dysfunction and greater disability.
Timed Up and Go Test | 24 Months
  The TUG test is a simple and effective measure of physical mobility, balance, and the risk of falls in individuals, especially those with Parkinson's Disease. It involves timing how long it takes a person to rise from a chair, walk 3 meters, turn around, walk back, and sit down again. The total time taken to complete the test is recorded in seconds.
  • Longer times suggest greater difficulty with mobility, balance, and overall motor function, which may indicate a higher fall risk and greater disability.
Parkinson's Disease Fatigue Scale (PFS-16) | 24 Months
  The PFS-16 is a self-reported tool that helps to assess the level of fatigue experienced by individuals with Parkinson's Disease. It consists of 16 questions that cover the frequency and impact of fatigue on daily life.
  • Scoring: Each item is rated on a scale from 1 to 5, where 1 = never and 5 = always. Total score range: 16 to 80

CONTACTS AND LOCATIONS:
Locations (2):
- Pakistan (2):
  - Chaudary Muhammad Akram Teaching Hospital, Azra Naheed Medical College, Superior University, Lahore, Punjab Province
  - Superior University CRC, Lahore, Punjab Province

IPD SHARING:
Plan to Share IPD: No